CLINICAL TRIAL: NCT02104154
Title: Evaluation of the Samsung LABGEO PT10 Hepatic Panel in a Point-of-Care Setting
Status: Terminated | Type: Observational
Why Stopped: To conduct interim analysis and assess whether assay changes are recommended.
Sponsor: Samsung Electronics (Industry)
Responsible Party: Sponsor
Other Study IDs: T10-02
Record Dates: First submitted 2013-12-13; First posted 2014-04-04 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Hepatic Disease
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Retaining serum and plasma specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- symptoms of liver disease: Device: Samsung LABGEO PT10 Hepatic Panel
  Interventions: Device: Samsung LABGEO PT10 Hepatic Panel

INTERVENTIONS:
Device: Samsung LABGEO PT10 Hepatic Panel

SUMMARY:
To establish the performance characteristics of the Samsung LABGEO PT10 by comparing the test results of the PT10 Hepatic assay with results obtained from an FDA-cleared chemistry analyzer.

DETAILED DESCRIPTION:
To establish the correlation between measurand values as obtained from the Samsung LABGEO PT10 Hepatic Panel at the point of care, and the corresponding measurand values as obtained on a commercial clinical chemistry analyzer, with respect to prospectively collected human serum specimens.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with a history of elevated liver enzymes or symptoms suggestive of elevated liver enzymes
* Presenting to the site and requiring testing for levels of liver enzymes as part of routine care at the site
* Subjects able and willing to provide written informed consent

Exclusion Criteria:

* Subjects unable or unwilling to provide written informed consent
* Subjects with a life-threatening disease or any serious, potentially life-threatening medical illness that may compromise patient safety or study conduct

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Bias between Samsung LABGEO PT10 serum results and matching FDA-cleared comparator assay | baseline

SECONDARY OUTCOMES:
Mean percentage difference between all pairs of plasma and serum measurements using Bland-Altman plot of differences. | baseline
Standard deviation and coefficients of variation of between run, between day and total precision. | 20 days
Estimates of reference intervals by computing the 2.5th percentile of associated distribution of test measurement (for each analyte) and the 97.5th percentile of associated distribution. | baseline
Mean percentage difference between all pairs of serum and whole blood measurements using Bland-Altman plot of differences. | baseline
Mean percentage difference between all pairs of plasma and whole blood measurements using Bland-Altman plot of differences. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nam Shin, Study Chair — Nexus DX
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States